CLINICAL TRIAL: NCT01508832
Title: Determination of the Duration of Action of a Lidocaine and a Bupivacaine Digital Nerve Block in Human Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 11-06121
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Onset and Duration of a Digital Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine 1% Digital Nerve Block (2 cc)
  Interventions: Drug: Lidocaine Digital Nerve Block
- Bupivacaine (Active Comparator): Bupivacaine 0.25% Digital Block (2 cc)
  Interventions: Drug: Bupivacaine Digital Block

INTERVENTIONS:
Drug: Lidocaine Digital Nerve Block — Lidocaine 1% Digital Nerve Block (2 cc
  Arms: Lidocaine
Drug: Bupivacaine Digital Block — Bupivacaine 0.25% Digital Block (2 cc)
  Arms: Bupivacaine

SUMMARY:
The duration of the autonomic (sympathetic) block will last longer than the sensory block. The duration of the increased perfusion index will last longer than either the sympathetic or sensory block.

DETAILED DESCRIPTION:
The Masimo SpHb™ (SpHb) is a device used to monitor the blood hemoglobin level via a sticky sensor connected to a finger. Our results from 2 recent studies undertaken with this device concluded: 1) that it is not always accurate when the finger is cold such as during surgical blood loss, and 2) a local nerve block to the finger improved the finger temperature and the accuracy of the device.

Our purpose is to investigate the duration of effect of two local nerve blocking drugs (lidocaine and bupivacaine - both FDA approved drugs in routine use) in a finger on each hand. Having a better understanding of how long the nerve block lasts could help determine when an additional block might be necessary to maintain the accuracy of the device during surgical blood loss.

We previously listed the primary outcome for this study as the time until return to baseline finger temperature. However, in blinded looks at the data it became clear that defining time until return to baseline from the serial temperature measurements in an objective fashion would be extremely difficult and potentially controversial. We have modified the primary outcome to be the change in the average temperature from baseline to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers

Exclusion Criteria:

* History of allergic response to local anesthetics
* BMI >25
* Pregnant of nursing
* Current smokers or past smokers of > 1 pack year history
* Neurological deficit and/or injury in the upper extremities
* Current respiratory infection
* Per investigator judgement, would not be suitable for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Miller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers recruited through local media source. Protocol consisted of a single study day in anesthesia research study space at the University of California San Francisco Parnassus campus.
Groups:
- Lidocaine Block, Right Finger; Bupivacaine Block, Left Finger: Lidocaine 1% digital nerve block (2cc), right finger; Bupivacaine 0.25% digital nerve block (2cc), left finger.
- Lidocaine Block, Left Finger; Bupivacaine Block, Right Finger: Lidocaine 1% digital nerve block (2cc), left finger; Bupivacaine 0.25% digital nerve block (2cc), right finger.
Period: Overall Study
Arm/Group | Lidocaine Block, Right Finger; Bupivacaine Block, Left Finger | Lidocaine Block, Left Finger; Bupivacaine Block, Right Finger
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine Block, Right Finger; Bupivacaine Block, Left Finger: Lidocaine 1% Digital Nerve Block (2 cc) , right finger. Bupivacaine 0.25% Digital Nerve Block (2 cc), left finger
- Lidocaine Block, Left Finger; Bupivacaine Block, Right Finger: Lidocaine 1% Digital Block (2cc), left finger; Bupivacaine 0.25% Digital Block (2 cc), right finger.
- Total: Total of all reporting groups
Arm/Group | Lidocaine Block, Right Finger; Bupivacaine Block, Left Finger | Lidocaine Block, Left Finger; Bupivacaine Block, Right Finger | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Average Finger Temperature From Baseline to Post-intervention.
Time Frame: 30 minutes prior and 240 minutes post intervention.
Population: The correspondingly-treated(lidocaine, bupivacaine) finger of all 12 study participants included in analysis for each arm/group
Measure: Mean (Standard Error); unit: degrees centigrade
Groups:
- Lidocaine: Lidocaine 1% digital nerve block (2cc) in one finger
- Bupivacaine: Bupivacaine 0.25% digital nerve block (2cc) in one finger
Arm/Group | Lidocaine | Bupivacaine
Number analyzed (Participants) | 12 | 12
degrees centigrade | -1.35 (0.71) | 0.93 (0.71)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Lidocaine: Lidocaine digital block in right or left finger
- Bupivacaine: Bupivacaine digital block right or left finger
Arm/Group | Lidocaine | Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=12) | Bupivacaine (N=12)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — 2-3 millimeter raised, reddened blister-like area at the base of both the right and left 4th finger of the same participant. No drainage, pain or irritation noted. Participant was contacted to verify resolution at 7 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No